CLINICAL TRIAL: NCT06218134
Title: Evaluate the Safety and Potential Efficacy of Human Wharton's Jelly-derived Mesenchymal Stem Cells (EN001) in Patients With Charcot-Marie-Tooth Disease Type 1E
Brief Title: Evaluate the Safety and Potential Efficacy of Human Wharton's Jelly-derived Mesenchymal Stem Cells With Charcot-Marie-Tooth Disease Type 1E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Byung-Ok Choi, MD, PhD, Professor, Department of Neurology, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2023-10-148
Record Dates: First submitted 2023-12-19; First posted 2024-01-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Charcot-Marie-Tooth Disease, Type 1
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- human Wharton's jelly-derived mesenchymal stem cells (EN001) (Experimental): * human Wharton's jelly-derived mesenchymal stem cells (EN001) dose of administration: 2.5x106 cells/kg
  * method of adminstration: one-time, intravenous administration
  Interventions: Biological: human Wharton's jelly-derived mesenchymal stem cells

INTERVENTIONS:
Biological: human Wharton's jelly-derived mesenchymal stem cells — human Wharton's jelly-derived mesenchymal stem cells(product name: EN001)

SUMMARY:
Charcot-Marie-Tooth disease (CMT) is a hereditary peripheral nerve disease that causes causes muscle atrophy, muscle weakness, sensory loss, balance disorder, gait disorder, blindness, hearing disorder, breathing disorder, vocal cord paralysis, foot deformity, scoliosis, and reflex dysfunction, More than 140 types of genes causing this disease are known. Charcot-Marie-Tooth (CMT) 1E, the target disease of this study, shows very severe symptoms compared to other Charcot-Marie-Tooth types. In cases of early onset, especially in children under 5 years of age, almost all patients are unable to walk without a wheelchair and have severe illness. Symptoms include scoliosis, breathing problems, vocal cord paralysis, foot deformity, loss of sensation and reflex function.

Additionally, more than 40% of Charcot-Marie-Tooth (CMT) 1E patients have hearing loss and become unable to live without hearing aids. Although this disease is very disabling, there is still no approved treatment.

To date, there is a lack of practical treatment or treatment support methods that can change the progression of hereditary motor and sensory neuropathy, so the focus is on pain control, use of assistive devices, and rehabilitation treatment, but the treatment effect is almost non-existent.

This study is conducted for the purpose of confirming the safety and exploratory treatment effect by administering EN001, an allogeneic umbilical cord-derived mesenchymal stem cell, once intravenously to patients with Charcot-Marie-Tooth (CMT) 1E.

EN001 is an allogeneic (alien-derived) umbilical cord-derived mesenchymal stem cell, and a phase 1 clinical trial of single intravenous administration was completed in 9 Charcot-Marie-Tooth (CMT) type 1A patients. Among the four adverse reactions that occurred in the participating research subjects, there were no adverse drug reactions related to EN001, and all four cases were mild and recovered. No serious adverse drug reactions or infusion reactions were observed in any study subjects, so this is a safe stem cell treatment.

Through efficacy tests and non-clinical tests, the effectiveness of improving behavior and increasing nerve and motor conduction speeds when administering the test drug to animal models of muscle disease was confirmed, so it is expected that this study can stabilize the disease progression in patients, and it will contribute to improving the quality of life and further promoting public health and welfare.

ELIGIBILITY:
Inclusion Criteria:

1. Those who voluntarily agreed to participate in this clinical study
2. Men and women over 19 years of age as of the date of written consent
3. Those who meet all of the following genetic and clinical diagnostic criteria

   * Genetic diagnosis: CMT1E

     * Clinical diagnosis

       * CMTNS score of 2 or more
       * Those with muscle weakness due to foot dorsiflexion
4. Women or men of childbearing potential who agreed to use the appropriate contraceptive method suggested in the protocol during the clinical study period.

   * Appropriate contraception is defined as follows, and is achieved by applying one or more methods of contraception.

     * Hormonal contraceptives
     * Implantation of an intrauterine device or intrauterine system
     * Sterilization procedures (vasectomy, tubal ligation, etc.)

Exclusion Criteria:

1. Those with the following comorbidities confirmed at the time of screening (1) Those who have a neuromuscular disease other than CMT1E or a neuropathy- causing factor (uremia) that may affect the safety and treatment effect of this clinical study, according to the judgment of the researcher. (2) Those diagnosed with type 1 or type 2 diabetes (3) Those diagnosed with active pulmonary tuberculosis (4) Patients with uncontrolled hypertension (systolic blood pressure over 180 mmHg or diastolic blood pressure over 110 mmHg) (5) Persons with other clinically significant diseases, including significant heart, lung, liver, kidney, hematological, immunological or behavioral diseases or malignant tumors, according to the judgment of the researcher. (6) Those who show the following test abnormalities in clinical laboratory tests at the time of screening

   * AST(spartate aminotransferase) or ALT(alanine aminotransferase) > 3 x ULN(upper limit of normal) ②Total bilirubin > 1.5 x ULN(upper limit of normal)

     * Serum creatinine > 1.5 x ULN(upper limit of normal)

       * D-dimer > 1.5 x ULN(upper limit of normal)

         ⑤ Serum virus test (HBsAg, anti-HBc, anti-HCV, Positive for any one of HIV Ag/Ab)

         - (If anti-HBc positive) However, registration is possible if the HBV DNA test result is negative.
         * (If anti-HCV positive) However, registration is possible if the HCV RNA test result is negative.
2. Medical history and surgical history

<!-- -->

1. Those who have undergone orthopedic surgery (bone or ligament correction, artificial joint implantation, osteotomy, arthroscopic surgery) on the lower extremities within 24 weeks before screening
2. Those with a history of stroke or cerebral ischemic attack within 48 weeks before screening
3. Those with a history of coronary artery disease, such as myocardial infarction or incomplete angina, within 48 weeks before screening
4. Persons with a history of malignant tumor within 240 weeks prior to screening (excluding basal cell carcinoma or squamous cell carcinoma that occurs on the skin) 3) Drugs and therapies prohibited from concurrent use

<!-- -->

1. A person who participated in another clinical trial and administered/applied an investigational drug or medical device within 4 weeks before screening
2. Those who administered/applied immunosuppressants, chemotherapy, radiation therapy, etc. within 12 weeks before screening
3. Those who administered stem cell therapy or gene therapy within 240 weeks before screening
4. Persons who have administered neurotoxic drugs that may accelerate peripheral nerve damage

   - Platinum series: cisplatin, carboplatin, oxaliplatin

   - Taxane series: paclitaxel, docetaxel

   - Proteasome inhibitors: bortezomib, carfilzomib, ixazomib, etc.

   - thalidomide and derivatives: thalidomide, lenalidomide, pomalidomide

   - Vinca alkaloid series: vincristine, vinblastine, vindesine, vinorelbine

   - Antiarrhythmic drug: amiodarone

   - Anti-inflammatory and antibiotic: colchicine, nitrofurantoin
   * Antiretroviral drugs: zalcitabine, stavudine
   * Others: dichloroacetate, tacrolimus, suramin 4) Persons with hypersensitivity to the components of human cells (EN001) used in this clinical study 5) Those who have had metal substances (heart pacemaker, nerve stimulator, cochlear implant, etc.) implanted in their body 6) Pregnant, lactating, or planning to become pregnant while participating in clinical research 7) Persons with a psychiatric disorder (anxiety disorder, claustrophobia, or other significant mental disorder) or a history of drug and alcohol abuse that may affect clinical research, according to the judgment of the researcher. 8) A person who is deemed inappropriate to participate in clinical research according to the judgment of the researcher.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Infusion-related reaction | up to 12month
  Check Fever, high blood pressure, low blood pressure, tachycardia, hyperventilation, rash, shock-related reactions related to administration

SECONDARY OUTCOMES:
Confirmation of exploratory treatment effect of jelly-derived mesenchymal stem cells(EN001) | up to 12month
  Charcot-Marie-Tooth disease 1E disease scale: CMTNS(Charcot-Marie-Tooth Neuropathy Score version 2), Lower values indicate better clinical conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- SMC, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No